CLINICAL TRIAL: NCT04082169
Title: Causes and Consequences of Primary Ovarian Insufficiency
Acronym: Clinical POI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2018/1206
Record Dates: First submitted 2019-08-20; First posted 2019-09-09 (Actual); Last update posted 2019-09-09 (Actual); Status verified 2019-08

CONDITIONS: Primary Ovarian Insufficiency; Premature Menopause
MeSH Terms: conditions — Primary Ovarian Insufficiency; Menopause, Premature

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — serum
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
100 women with primary ovarian insufficiency will be included for extensive diagnostic workup to improve diagnostic precision by extended autoantibody screening and genetic and toxicological testing.

ELIGIBILITY:
Inclusion Criteria:Women 40 years or younger, more than 4 months amenorrhea, more than 2 FSH measurements in menopausal range (drawn at least 2 months apart), ability to provide informed concent -

Exclusion Criteria:History of oophorectomy, chemotherapy or radiation

-

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Ovarian insufficiency
Study Population: 100 women with primary ovarian insufficiency defined as absence of menstruation more than 4 months and serum level of follicle stimulation hormone (FSH) in menopausal range at 2 or more occations
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-01-11 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Autoimmune | one day
  Prevalence of primary ovarian insufficiency (POI) with autoimmune etiology based on positive autoantibodies toward steroidogenic cells
Genetic | one day
  Prevalence of POI with genetic etiology defined by detection of genetic defects in a NGS panel
Endocrine disrupting chemicals | one day
  Characterize the cohort of women with POI, including testing for environmental factors

SECONDARY OUTCOMES:
Phenotype description | one day
  Describe phenotypical characteristics including menstrual characteristics, hormone profile, BMD

CONTACTS AND LOCATIONS:
Overall Officials: Kahtan Al-Azawy, MD, Study Chair — Haukeland University Hospital
Locations (1):
- HaukelandUH, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vogt EC, Bratland E, Berland S, Berentsen R, Lund A, Bjornsdottir S, Husebye E, Oksnes M. Improving diagnostic precision in primary ovarian insufficiency using comprehensive genetic and autoantibody testing. Hum Reprod. 2024 Jan 5;39(1):177-189. doi: 10.1093/humrep/dead233. PMID 37953503